CLINICAL TRIAL: NCT04155151
Title: Feasibility Study to Assess if Using the 6 Minute Walk Test at a Patients First Visit to Surgical Outpatients Will Identify Those Individuals With a Significantly Reduced Level of Cardiorespiratory Fitness.
Brief Title: Can the 6MWT Can be Used to Identify Reduced Patient Fitness at Surgical Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STH21039
Record Dates: First submitted 2019-10-29; First posted 2019-11-07 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Surgery

STUDY DESIGN:
Intervention Model Description: Prospective observational
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): 6 Minute Walking Test
  Interventions: Other: 6 minute walk test

INTERVENTIONS:
Other: 6 minute walk test — A test of fitness that requests the participant to walk as far as they can at their own pace in 6 minutes, the distance walked in those 6 minutes is recorded.

SUMMARY:
The aim of this study is to assess the feasibility of using the 6 minute walk test (6MWT) as a cardiorespiratory fitness (CRF) screening tool. The screening would take place when the patient attends the hospital for their initial surgical outpatient appointment. By screening all potential major intra-abdominal surgery patients for a period of 6 months and recording the distance walked in the 6 minutes (6MWD) the aim is to produce a threshold distance for the patients of Sheffield that would identify those with sufficient CRF what would allow them to proceed to surgery without further investigations or fitness interventions.

Having identified the fit it would allow the perioperative team to focus resources on the less fit with the aim of improving CRF and other elements that would lead to reduced postoperative morbidity and mortality.

Other primary aims include noting the time to surgery. This data will inform on wither instigation of the early screening test would facilitate enrolment and completion of an exercise programme before surgery.

The secondary aim is to assess the relationship between the 6MWD and routine CPET to confirm if those that walk the furthest are in fact the fittest.

DETAILED DESCRIPTION:
This is a prospective observational study that would run for a period of 6 months. The population proceeding to undergo major abdominal surgery is estimated to be 500 patients a year. The primary aim is to invite all patients being considered for major abdominal surgery to participate in a simple screening test of fitness, the 6 minute walk test (6MWT).

Potential participants would be identified by the participating surgical teams during their first visit to this institutions Surgical Outpatient Department (SOPD). Upon identification the individual would be provided with information designed to be read on returning to the waiting area from the SOPD clinic room.

The study walker, who would be an appropriately trained research nurse or outpatient clinic support worker, would approach the patient to answer questions and provide further information if required. Consent for participation would then be obtained. The participating individual would then be walked the short distance to the testing area and would be offered a seat whilst the 6MWT procedure was explained in more detail. Time would be allowed for questions. The 6MWT would be then conducted as per the American Thoracic Society guidance. Heart rate will be recorded manually both at baseline and at the cessation of the test.

Following the 6MWT patients could either depart the hospital or return to the SOPD if it was felt a period of recovery was required.

The 6 minute walk distance (6MWD) would be recorded against the patient's participant study identification number. Patient identifiers that would link the patient study number to a particular patient would be stored safely behind lock and key or encryption when electronic. The case report forms will be paper to allow timely collection of data and this information will be collated onto a spreadsheet which will facilitate future analysis.

At a later date information will also be collected on date of operation, this will be used to assess the present 'window' of opportunity for enrolling the less fit into an exercise programme.

A secondary aim of this study is to investigate the relationship between the 6MWD and the objectively measured anaerobic threshold and peak oxygen consumption that will be obtained when some of these patients undergo cardiopulmonary exercise testing (CPET) as part of their standard pathway to surgery. Reports produced following CPET interpretation are stored as PDFs upon this institutions server, named individuals involved in collecting data for this study will have access to the this server to complete case report forms that require details from the CPET reports.

Statistical analysis:

Descriptive statistics will be undertaken on the population that participates in the 6MWT, the population will be split into quartiles based on what the investigators know about our non-cardiopulmonary surgery population following analysis of our CPET database. Those deemed significantly less fit occupied the lowest quartile. The aim would be to assess for population normality and produce thresholds for the most fit; the greatest distance walked by 25% of the population with the least fit the lowest 25% of the population. The middle 50% would be less fit.

Linear regression analysis will be used to determine the 6MWD threshold that correlates with a level of anaerobic threshold or peak oxygen consumption objectively measured by CPET, deemed acceptable and indicating those individuals for whom no further preoperative interventions are required.

During the 12 months of 2017 the investigators undertook 483 preoperative major abdominal surgery cardiopulmonary exercise (CPET) tests. The investigators anticipate collecting 6MWT data on 250 patients and CPET data on at least 240 patients. Hopefully all those who undergo CPET will have consented to undergo a 6MWT whilst in the SOPD during their first visit on their pathway toward surgery.

ELIGIBILITY:
Inclusion Criteria:

* Considered for major abdominal surgery who can weight bear

Exclusion Criteria:

* Considered for major surgery who cannot weight bear
* Unable to follow the verbal instructions on walking test procedure provided by the researcher

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Can all the patients invited to 6MWT complete the walk test | Day 1
  Number of participants who are able to complete the walk test at their first visit
Distance walked by the participants during the 6MWT measured in meters | Day 1
  measured in meters completed
The duration in time between the walk test and the participant attending for surgery | within 60 days of original single point measurement
  measured in days

SECONDARY OUTCOMES:
Correlation between the distance walked during the 6 minute walk test and anaerobic threshold as measured by cardiopulmonary exercise testing (CPET) in ml/kg/min. | for 90 days beyond the closure of the study
  statistical analysis
Correlation between the distance walked during the 6 minute walk test and peak oxygen consumption as measured by cardiopulmonary exercise testing (CPET) in ml/kg/min. | for 90 days beyond the closure of the study
  statistical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Angela Pinder, Study Chair — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Northern General Hospital, Sheffield, South Yorks, United Kingdom

IPD SHARING:
Plan to Share IPD: No